CLINICAL TRIAL: NCT00547898
Title: Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Two-Stage Study to Assess the Efficacy and Safety of 3 Doses of Crofelemer Orally Twice Daily for the Treatment of HIV-Associated Diarrhea
Brief Title: Safety and Effectiveness of 3 Doses of Crofelemer Compared to Placebo in the Treatment of HIV Associated Diarrhea
Acronym: ADVENT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP303-101
Record Dates: First submitted 2007-10-21; First posted 2007-10-23 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: HIV Associated Diarrhea
Keywords: HIV; AIDS; Diarrhea; HIV Associated Diarrhea
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Diarrhea | interventions — crofelemer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Experimental)
  Interventions: Drug: Placebo
- Crofelemer 125 mg (Experimental)
  Interventions: Drug: Crofelemer 125 mg
- Crofelemer 250 mg (Experimental)
  Interventions: Drug: Crofelemer 250 mg
- Crofelemer 500 mg (Experimental)
  Interventions: Drug: Crofelemer 500 mg

INTERVENTIONS:
Drug: Crofelemer 125 mg — Crofelemer 125 mg
  Arms: Crofelemer 125 mg
Drug: Crofelemer 250 mg — Crofelemer 250 mg
  Arms: Crofelemer 250 mg
Drug: Crofelemer 500 mg — Crofelemer 500 mg
  Arms: Crofelemer 500 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, parallel-group, placebo-controlled, multi-center study. This study will compare an investigational new drug (crofelemer) to placebo for the control of HIV-associated diarrhea. The first stage of the study will determine the optimal dose of study drug based on safety and response to therapy and the second stage will evaluate further the effectiveness of the optimal dose.

ELIGIBILITY:
Inclusion Criteria:

* History of HIV-1 infection confirmed by standard serological tests
* Stable medical regimen for treatment of HIV disease and associated conditions for at least 4 weeks prior to screening
* Patient-reported history of diarrhea, defined as either persistently loose stools despite regular ADM use, or one or more watery bowel movements per day without regular ADM use, of at least 1 month duration
* Colonoscopy within the past 5 years if ≥ 50 years of age.

Exclusion Criteria:

* Pregnancy or breast-feeding
* Current or past gastrointestinal (GI) medical or surgical conditions
* Use of certain opiate pain medication within 2 weeks of screening
* Use of an antibiotic within 2 weeks prior to screening, with the exception of stable antibiotic therapy for prophylactic treatment of infection or an HIV-associated condition
* CD4 counts < 100 cells/mm3
* Previous randomization into this study, or into any other crofelemer study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2007-10; Primary Completion 2011-01-27 (Actual); Study Completion 2011-07-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (59):
- United States (56):
  - Huntsville, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Bakersfield, California
  - Beverly Hills, California
  - Fountain Valley, California
  - Long Beach, California
  - Los Angeles, California
  - Oakland, California
  - Palm Springs, California
  - San Diego, California
  - San Francisco, California
  - San Mateo, California
  - Denver, Colorado
  - Daytona Beach, Florida
  - Fort Lauderdale, Florida
  - Ft. Pierce, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Orlando, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Wilton Manors, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Iowa City, Iowa
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - Santa Fe, New Mexico
  - Great Neck, New York
  - Manhasset, New York
  - Mount Vernon, New York
  - New York, New York
  - Rochester, New York
  - The Bronx, New York
  - Gastonia, North Carolina
  - Cincinnati, Ohio
  - Portland, Oregon
  - Columbia, South Carolina
  - Austin, Texas
  - Bellaire, Texas
  - Dallas, Texas
  - Harlingen, Texas
  - Houston, Texas
  - Longview, Texas
  - San Antonio, Texas
  - Lynchburg, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Spokane, Washington
- Puerto Rico (3):
  - Ponce
  - Rio Piedras
  - San Juan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Crofelemer 125 mg | Crofelemer 250 mg | Crofelemer 500 mg
Started | 138 | 136 | 54 | 46
Completed | 129 | 126 | 54 | 40
Not Completed | 9 | 10 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Crofelemer 125 mg | Crofelemer 250 mg | Crofelemer 500 mg | Total
Number analyzed (Participants) | 138 | 136 | 54 | 46 | 374
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (8.42) | 45 (7.66) | 43.8 (8.37) | 45.8 (9.06) | 44.9 (1.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 6 | 7 | 56
  Male | 116 | 115 | 48 | 39 | 318

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Outcome is Count of Participants With Two or Less Watery Bowel Movements Per Week During at Least Two Weeks of the Treatment Phase of the Optimal Dose of Crofelemer Compared to Placebo
Time Frame: 31 days
Population: The primary efficacy analysis was pre-specified to be for the optimal dose of crofelemer compared to placebo. Crofelemer 125 mg BID group was selected as the optimal dose. Since other doses of crofelemer were not considered to be the optimal dose, they are not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Crofelemer 125Mg BID | Placebo BID
Number analyzed (Participants) | 136 | 138
Participants | 24 | 11

2. Other Pre Specified Outcome: Percentage of Participants Experiencing Relief of Diarrhea
Description: Relief of diarrhea was defined as two or less watery bowel movements per week during at least two weeks of the treatment phase.
Time Frame: 31 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Crofelemer 125 mg | Crofelemer 250 mg | Crofelemer 500 mg
Number analyzed (Participants) | 138 | 136 | 54 | 46
Participants | 11 | 24 | 5 | 9

ADVERSE EVENTS:
Description: The safety population included participants who received study drug and had at least one post baseline assessment. The safety population was comprised of 226 crofelemer particpants and 137 placebo participants.
Arm/Group | Placebo | Crofelemer 125 mg | Crofelemer 250 mg | Crofelemer 500 mg
Serious Adverse Events (participants affected / at risk) | 4/137 | 2/130 | 0/54 | 0/42
Other Adverse Events (participants affected / at risk) | 0/137 | 0/130 | 0/54 | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=137) | Crofelemer 125 mg (N=130) | Crofelemer 250 mg (N=54) | Crofelemer 500 mg (N=42)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 0 | 0 | 0
ESCHERICHIA SEPSIS (Infections and infestations) | 0 | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 1 | 1 | 0 | 0
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes